CLINICAL TRIAL: NCT02385799
Title: A Controlled Trial of Sertraline in Young Children With Autism Spectrum Disorder
Brief Title: A Trial of Sertraline in Young Children With Autism Spectrum Disorder
Acronym: Sert2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Randi J. Hagerman, MD (Other)
Collaborators: Health Resources and Services Administration (HRSA) (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, Randi J. Hagerman, MD, UC Davis MIND Institute Medical Director, University of California, Davis
Organization: University of California, Davis (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 663866
Record Dates: First submitted 2015-02-09; First posted 2015-03-11 (Estimated); Results first posted 2019-05-09 (Actual); Last update posted 2019-10-22 (Actual); Status verified 2019-10

CONDITIONS: Autism Spectrum Disorder
Keywords: Autism Spectrum Disorder; Behavior; sertraline; treatment
MeSH Terms: conditions — Autism Spectrum Disorder; Behavior | interventions — Sertraline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sertraline Liquid Placebo (Placebo Comparator): The placebo will be dosed in an age depended manner. Participants aged 2-3 years of age will be given 2.5 mg of liquid placebo once per day for a period of six months. Participants aged 4 years to 6 years will be given 5 mg of liquid placebo once per day for a period of six months.
  Interventions: Drug: Sertraline Liquid Placebo
- Sertraline Active Medication (Active Comparator): Liquid sertraline (20 mg/cc) will be dosed in an age depended manner. Participants aged 2-3 years of age will be given 2.5 mg of liquid sertraline once per day for a period of six months. Participants aged 4 years to 6 years will be given 5 mg of liquid sertraline once per day for a period of six months.
  Interventions: Drug: Sertraline

INTERVENTIONS:
Drug: Sertraline Liquid Placebo — Liquid placebo given in parallel to active medication
  Other Names: Placebo
  Arms: Sertraline Liquid Placebo
Drug: Sertraline — Active medication
  Other Names: Zoloft
  Arms: Sertraline Active Medication

SUMMARY:
This study is a control trial of sertraline (Zoloft) in children aged 2 to 5 years old inclusive with Autism Spectrum Disorder. The trial is six months long, and each participant will receive a series of tests at both the beginning and end of the study. The researchers hope to show improvements in language and social deficits.

DETAILED DESCRIPTION:
This is a single center study and the UC Davis MIND Institute for Autism Spectrum Disorder (ASD) patients aged between 2 years and 5 years old inclusive funded by the Health Resources and Services Administration (HRSA). It is a double-blind control trial of sertraline (Zoloft), an anti-depressant typically used in the treatment of depression, obsessive-compulsive disorder, panic disorder, and other conditions. The researchers are investigating the use of this selective serotonin reuptake inhibitor (SSRI) in ASD because a retrospective study has shown significant improvements in language and social deficits. There is also emerging evidence regarding the stimulation of brain-derived neurotrophic factor (BDNF) and the stimulation of neurogenesis when an SSRI is given early on in the development of animal models of Down syndrome. The researchers hope to see improvements in language stimulation, social gaze and social reciprocity, spatial attention, and a decrease in autistic behaviors.

The aim of this study is to carry out a double-blind placebo controlled trial of sertraline in children with ASD who are between the ages of 2 years and 5 years old inclusive. At baseline, the researchers will assess behavioral and cognitive development. Each participant will be involved in this trial for a period of six months. This will include three visits to the UC Davis MIND Institute and eight phone calls. The researchers will also assess the side effects of the sertraline treatment throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Documentation of Autism Spectrum Disorder with Diagnostic and Statistical Manual for Mental Disorders-Fifth edition, criteria as well as a standardized autism assessment such as the Autism Diagnostic Observation Schedule or the Autism Diagnostic Interview-Revised.
* Subject between the ages of 24-72 months of age.
* A reliable parent or caregiver who can report the side effects and communicate effectively with the research team.
* Stable medications during the two months prior to enrollment.
* Currently receiving interventions in the community or school for Autism Spectrum Disorder

Exclusion Criteria:

* Current or past Selective Serotonin Reuptake Inhibitor treatment.
* Other serious co-morbid medical disorders affecting brain function and behavior, including uncontrolled seizures.

Ages: 24 Months to 72 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 58 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Randi J Hagerman, M.D., Principal Investigator — UC Davis MIND Institute
Locations (1):
- UC Davis MIND Institute, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Potter LA, Scholze DA, Biag HMB, Schneider A, Chen Y, Nguyen DV, Rajaratnam A, Rivera SM, Dwyer PS, Tassone F, Al Olaby RR, Choudhary NS, Salcedo-Arellano MJ, Hagerman RJ. A Randomized Controlled Trial of Sertraline in Young Children With Autism Spectrum Disorder. Front Psychiatry. 2019 Nov 6;10:810. doi: 10.3389/fpsyt.2019.00810. eCollection 2019. PMID 31780970

RESULTS

PARTICIPANT FLOW:
Groups:
- Sertraline Liquid Placebo: The placebo will be dosed in an age depended manner. Participants aged 2-3 years of age at enrollment will be given 2.5 mg of liquid placebo once per day for a period of six months. Participants aged 4-5 years at enrollment will be given 5 mg of liquid placebo once per day for a period of six months.
  Sertraline Liquid Placebo: Liquid placebo given in parallel to active medication
- Sertraline Active Medication: Liquid sertraline (20 mg/cc) will be dosed in an age depended manner. Participants aged 2-3 years of age at enrollment will be given 2.5 mg of liquid sertraline once per day for a period of six months. Participants aged 4-5 years at enrollment will be given 5 mg of liquid sertraline once per day for a period of six months.
  Sertraline: Active medication
Period: Overall Study
Arm/Group | Sertraline Liquid Placebo | Sertraline Active Medication
Started | 26 | 32
Completed End-of-Treatment Visit (Includes all subjects who returned for end-of-treatment study visit, including early terminations.) | 21 | 26
Completed (Includes all subjects who completed 6-month treatment with study drug. Excludes early terminations.) | 21 | 24
Not Completed | 5 | 8
Not completed — Lost to Follow-up | 1 | 2
Not completed — Adverse Event | 4 | 2
Not completed — Withdrawal by Subject | 0 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sertraline Liquid Placebo | Sertraline Active Medication | Total
Number analyzed (Participants) | 26 | 32 | 58
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 26 | 32 | 58
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 3.70 (1.10) | 4.31 (0.90) | 4.005 (1.00)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 7 | 12
  Male | 21 | 25 | 46
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 3 | 11
  Not Hispanic or Latino | 18 | 29 | 47
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 7 | 11
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 5 | 7
  White | 18 | 19 | 37
  More than one race | 2 | 1 | 3
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 26 | 32 | 58
The Autism Diagnostic Observation Schedule-Second Edition (ADOS-2) [Mean (Standard Deviation); unit: units on a scale] — The Autism Diagnostic Observation Schedule-Second Edition (ADOS-2) The assessment will provide a continuous metric of autism symptom severity for use in characterizing the participant sample and as a potential moderator of treatment response. The ADOS is a gold-standard measure of current symptoms of autism. Total scores will be used to assign a severity score. Scores range from 1 to 10, with higher scores reflecting more severe impairment
  units on a scale | 7.88 (1.62) | 7.34 (1.58) | 7.58 (1.60)

OUTCOME MEASURES:

1. Primary Outcome: Change in Mullen Scales of Early Learning - Expressive Language Raw Score
Description: The Mullen Scales of Early Learning (MSEL) is a cognitive test to measure cognitive ability and language development. The test has five scales: gross motor, visual reception, fine motor, receptive language, and expressive language. Shown here are the baseline and 6-month follow-up raw scores from the expressive language scale. This scale's raw scores range from 0 to 50. The lower the score on this scale, the weaker the ability; the higher the score, the greater the ability. The MSEL was administered at the baseline visit and at the 6-month follow-up visit.
Time Frame: From baseline visit to six-month visit
Population: Placebo group: 5 discontinued treatment, 0 of whom returned to complete follow-up assessments, so 21 subjects were analyzed at follow-up. Sertraline group: 8 discontinued treatment, 2 of whom returned voluntarily to complete follow-up assessments, so 26 subjects were analyzed at follow-up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sertraline Liquid Placebo | Sertraline Active Medication
Number analyzed (Participants) | 26 | 32
score on a scale
  Baseline | 19.69 (11.69) | 18.19 (10.39)
  Follow-up: number analyzed (Participants) | 21 | 26
  Follow-up | 21.81 (14.29) | 20.31 (11.70)

2. Primary Outcome: Change in Mullen Scales of Early Learning - Combined Age Equivalent Score
Description: The Mullen Scales of Early Learning (MSEL) is a cognitive test to measure cognitive ability and language development. The test has five scales: gross motor, visual reception, fine motor, receptive language, and expressive language. Shown here are the baseline and 6-month follow-up combined age equivalent scores, calculated as the sum of the age equivalent scores from each scale. The combined score ranges from 0 to 280. The lower the score on this scale, the weaker the ability; the higher the score, the greater the ability. The MSEL was administered at the baseline visit and at the 6-month follow-up visit.
Time Frame: From baseline visit to six-month visit
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sertraline Liquid Placebo | Sertraline Active Medication
Number analyzed (Participants) | 26 | 32
score on a scale
  Baseline | 25.61 (11.73) | 24.98 (12.79)
  Follow-up: number analyzed (Participants) | 21 | 26
  Follow-up | 30.30 (15.58) | 28.16 (14.15)

3. Secondary Outcome: Vineland Adaptive Behavior Scales, Second Edition (Vineland-II) Adaptive Behavior Composite Standard Score
Description: The Vineland-II measures the personal and social skills of individuals from birth through adulthood. It was designed to assess handicapped and non-handicapped persons in their personal and social functioning and is appropriate for individuals of all ages. The Vineland-II is a survey that is administered to a parent or caregiver using a semi-structured interview format and is organized around four Behavior Domains: Communication, Daily Living Skills, Socialization, and Motor Skills. Each subtest is scored with a standard score X=100 ± 15 and summed to calculate the Adaptive Behavior Composite (ABC) using age-adjusted scoring tables. Reported here are the ABC mean standard scores for the placebo and treatment groups at baseline. The ABC ranges from 20 to 160 and indicates low (20-70), moderately low (70-85), adequate (85-115), moderately high (115-130), or high (130-160) overall adaptive functioning.
Time Frame: At baseline visit
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sertraline Liquid Placebo | Sertraline Active Medication
Number analyzed (Participants) | 26 | 32
score on a scale | 68.50 (11.14) | 60.03 (12.15)

4. Secondary Outcome: Vineland Adaptive Behavior Scales, Second Edition (Vineland-II) Adaptive Behavior Composite Standard Score
Description: The Vineland-II measures the personal and social skills of individuals from birth through adulthood. It was designed to assess handicapped and non-handicapped persons in their personal and social functioning and is appropriate for individuals of all ages. The Vineland-II is a survey that is administered to a parent or caregiver using a semi-structured interview format and is organized around four Behavior Domains: Communication, Daily Living Skills, Socialization, and Motor Skills. Each subtest is scored with a standard score X=100 ± 15 and summed to calculate the Adaptive Behavior Composite (ABC) using age-adjusted scoring tables. Reported here are the ABC mean standard scores for the placebo and treatment groups at the six-month visit. The ABC ranges from 20 to 160 and indicates low (20-70), moderately low (70-85), adequate (85-115), moderately high (115-130), or high (130-160) overall adaptive functioning.
Time Frame: At six-month visit
Population: Placebo group: 5 discontinued treatment, 0 of whom returned to complete follow-up assessments, so 21 subjects were analyzed at follow-up. Sertraline group: 8 discontinued treatment, 2 of whom returned for an end-of-treatment visit, but due to time limitations only 1 of these 2 completed this assessment, so 25 subjects were analyzed at follow-up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sertraline Liquid Placebo | Sertraline Active Medication
Number analyzed (Participants) | 21 | 25
score on a scale | 71.52 (15.47) | 69.68 (15.14)

5. Secondary Outcome: Preschool Anxiety Scale-Revised - Total Score
Description: Preschool Anxiety Scale-Revised (PAS-R) is a questionnaire designed to assess symptoms of anxiety and fears in young children aged 6 and below as reported by their parents. The PAS-R consists of 34 questions, each with a rating option of 0 to 4 where 0=not true at all, 1=seldom true, 2=sometimes true, 3=quite often true, and 4=very often true. The total score is calculated as the sum of all responses and therefore ranges from 0 to 136. Lower scores indicate less anxiety/fear; higher scores indicate more anxiety/fear. Reported here are the mean total scores for the placebo and treatment groups at baseline.
Time Frame: At baseline visit
Population: Placebo group: staff inadvertently neglected to administer this questionnaire to the 2 subjects' caregivers at baseline, so only 24 were completed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sertraline Liquid Placebo | Sertraline Active Medication
Number analyzed (Participants) | 24 | 32
score on a scale | 15.38 (12.51) | 14.75 (11.58)

6. Secondary Outcome: Preschool Anxiety Scale-Revised - Total Score
Description: Preschool Anxiety Scale-Revised (PAS-R) is a questionnaire designed to assess symptoms of anxiety and fears in young children aged 6 and below as reported by their parents. The PAS-R consists of 34 questions, each with a rating option of 0 to 4 where 0=not true at all, 1=seldom true, 2=sometimes true, 3=quite often true, and 4=very often true. The total score is calculated as the sum of all responses and therefore ranges from 0 to 136. Lower scores indicate less anxiety/fear; higher scores indicate more anxiety/fear. Reported here are the mean total scores for the placebo and treatment groups at the six-month visit.
Time Frame: At six-month visit
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sertraline Liquid Placebo | Sertraline Active Medication
Number analyzed (Participants) | 21 | 26
score on a scale | 11.43 (10.04) | 14.77 (14.45)

7. Secondary Outcome: Preschool Language Scale-Fifth Edition - Total Language Raw Score
Description: The Preschool Language Scale-Fifth Edition (PLS-5) is designed to measure auditory comprehension (AC) and expressive communication (EC) for children from birth to 7 years 11 months. The measure examines the child's attention, play, gestures, social communication, semantics, language structure, integrative language skills and emergent literacy skills. The PLS-5 has expanded coverage of early play behaviors, concepts, theory of mind, and emergent literacy skills. The PLS-5 yields norm-referenced scores including standard scores, percentile ranks and age equivalents for the AC and EC scales as well as for Total Language (TL). Raw score ranges are 0 to 65 in AC, 0 to 67 in EC, and therefore 0 to 132 in TL (calculated by summing AC+EC raw scores). The higher the scores, the greater the language ability. Shown here are the mean TL raw scores from the baseline visit.
Time Frame: At baseline visit
Population: Sertraline group: 2 subjects were completely nonverbal at baseline, so the rater determined that their assessments could not be completed; therefore, only 30 subjects in this arm were analyzed at baseline.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sertraline Liquid Placebo | Sertraline Active Medication
Number analyzed (Participants) | 26 | 30
score on a scale | 48.65 (25.57) | 43.03 (23.35)

8. Secondary Outcome: Preschool Language Scale-Fifth Edition - Total Language Raw Score
Description: The Preschool Language Scale-Fifth Edition (PLS-5) is designed to measure auditory comprehension (AC) and expressive communication (EC) for children from birth to 7 years 11 months. The measure examines the child's attention, play, gestures, social communication, semantics, language structure, integrative language skills and emergent literacy skills. The PLS-5 has expanded coverage of early play behaviors, concepts, theory of mind, and emergent literacy skills. The PLS-5 yields norm-referenced scores including standard scores, percentile ranks and age equivalents for the AC and EC scales as well as for Total Language (TL). Raw score ranges are 0 to 65 in AC, 0 to 67 in EC, and therefore 0 to 132 in TL (calculated by summing AC+EC raw scores). The higher the scores, the greater the language ability. Shown here are the mean TL raw scores from the six-month visit.
Time Frame: At six-month visit
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sertraline Liquid Placebo | Sertraline Active Medication
Number analyzed (Participants) | 21 | 25
score on a scale | 57.24 (26.26) | 51.40 (23.56)

9. Secondary Outcome: Sensory Processing Measure-Preschool - Social Participation Raw Score
Description: The Sensory Processing Measure-Preschool (SPM-P) is a questionnaire measuring specific problems, including under- and over-responsiveness, sensory-seeking behavior, and perceptual problems in multiple environments (at home, at school, and in the community) for children aged 2 to 5 years old, as reported by the parent/caregiver. The SPM-P provides norm-referenced standard scores for two higher-level integrative functions (praxis and social participation) and five sensor sensory systems (visual, auditory, tactile, proprioceptive, and vestibular functioning). Reported here is the Social Participation subscale mean raw score at baseline, which ranges from 8 to 32. The lower the raw score, the more limited the child's level of social participation. The higher the score, the greater the child's level of social participation.
Time Frame: At baseline visit
Population: Placebo group: staff inadvertently neglected to administer this questionnaire to 1 subject's caregiver at baseline, so only 25 were completed. Sertraline group: staff inadvertently neglected to administer this questionnaire to 1 subject's caregiver at baseline, so only 31 were completed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sertraline Liquid Placebo | Sertraline Active Medication
Number analyzed (Participants) | 25 | 31
score on a scale | 21.96 (3.81) | 22.39 (5.10)

10. Secondary Outcome: Sensory Processing Measure-Preschool - Social Participation Raw Score
Description: The Sensory Processing Measure-Preschool (SPM-P) is a questionnaire measuring specific problems, including under- and over-responsiveness, sensory-seeking behavior, and perceptual problems in multiple environments (at home, at school, and in the community) for children aged 2 to 5 years old, as reported by the parent/caregiver. The SPM-P provides norm-referenced standard scores for two higher-level integrative functions (praxis and social participation) and five sensor sensory systems (visual, auditory, tactile, proprioceptive, and vestibular functioning). Reported here is the Social Participation subscale mean raw score at the six-month visit, which ranges from 8 to 32. The lower the raw score, the more limited the child's level of social participation. The higher the score, the greater the child's level of social participation.
Time Frame: At six-month visit
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sertraline Liquid Placebo | Sertraline Active Medication
Number analyzed (Participants) | 21 | 25
score on a scale | 20.86 (4.07) | 21.16 (5.04)

11. Secondary Outcome: Clinical Global Impression Scale-Severity (CGI-S)
Description: The Clinical Global Impression-Severity (CGI-S) is a 7-point scale completed by a clinician that yields a rating of the patient's illness severity at the time of assessment, relative to the clinician's past experience with patients who have the same diagnosis. The 7-point scale ranges from: 1 = Normal; 2 = Borderline Ill; 3 = Mildly Ill; 4 = Moderately Ill; 5 = Markedly Ill; 6 = Severely Ill; and 7 = Extremely Ill. Therefore, the higher the score, the greater the severity of the patient's illness. The CGI-S was administered at baseline only for the purpose of characterizing the study population. Shown here are the CGI-S mean scores from the baseline visit.
Time Frame: At baseline visit
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sertraline Liquid Placebo | Sertraline Active Medication
Number analyzed (Participants) | 26 | 32
score on a scale | 4.38 (0.98) | 4.66 (0.94)

12. Secondary Outcome: Clinical Global Impression Scale-Improvement (CGI-I)
Description: The Clinical Global Impression-Improvement (CGI-I) is a 7-point scale completed by a clinician that yields a score measuring the overall behavioral change of an individual and their therapeutic response. The 7-point scale ranges from: 1 = Very much improved; 2 = Much improved; 3 = Minimally improved; 4 = No change; 5 = Minimally worse; 6 = Much worse; and 7 = Very much worse. Therefore, the lower the score, the greater the behavioral improvement as rated by the clinician. The CGI-I was administered at the three-month and six-month visits. Shown here are the CGI-I mean scores from the 3-month follow-up visit.
Time Frame: At three-month visit
Population: Placebo group: 3 discontinued treatment/become lost to follow-up prior to reaching 3-month visit, so 23 subjects were analyzed at this timepoint. Sertraline group: 5 discontinued treatment/become lost to follow-up prior to reaching 3-month visit, so 27 subjects were analyzed at this timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sertraline Liquid Placebo | Sertraline Active Medication
Number analyzed (Participants) | 23 | 27
score on a scale | 2.65 (1.11) | 2.70 (1.03)

13. Secondary Outcome: Clinical Global Impression Scale-Improvement (CGI-I)
Description: The Clinical Global Impression-Improvement (CGI-I) is a 7-point scale completed by a clinician that yields a score measuring the overall behavioral change of an individual and their therapeutic response. The 7-point scale ranges from: 1 = Very much improved; 2 = Much improved; 3 = Minimally improved; 4 = No change; 5 = Minimally worse; 6 = Much worse; and 7 = Very much worse. Therefore, the lower the score, the greater the behavioral improvement as rated by the clinician. The CGI-I was administered at the three-month and six-month visits. Shown here are the CGI-I mean scores from the 6-month follow-up visit.
Time Frame: At six-month visit
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sertraline Liquid Placebo | Sertraline Active Medication
Number analyzed (Participants) | 21 | 26
score on a scale | 1.14 (0.96) | 1.23 (1.11)

14. Secondary Outcome: Visual Analog Scale - Language/Communication Score
Description: The Visual Analog Scale measures the severity of three specific behavioral symptoms as reported by the parent/caregiver: Language/Communication, Anxiety/Obsessive Compulsive Behaviors, and Aggression/Hyperactivity/Hyperarousal. Caregivers mark on a visual line measuring 10 cm with "worst behavior" at 0 cm and "best behavior" at 10 cm. For each behavior the caregiver is instructed to mark their impression of the behavior at baseline visit and again at the six-month visit. The calculated distance in cm between the marks drawn at the baseline and six-month visits thereby demonstrates whether each behavior improved, worsened, or stayed the same during the study, and by how much. Shown here is the mean distance in cm from the "worst behavior" side for the Language/Communication scale, at baseline. The smaller the value, the worse the behavior. The range is minimum 0 cm to maximum 10 cm.
Time Frame: At baseline visit
Population: Placebo group: staff inadvertently neglected to administer this assessment to 1 subject's caregiver at baseline, so only 25 were completed. Sertraline group: staff inadvertently neglected to administer this assessment to 1 subject's caregiver at baseline, so only 31 were completed.
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | Sertraline Liquid Placebo | Sertraline Active Medication
Number analyzed (Participants) | 25 | 31
centimeters | 2.84 (2.04) | 2.03 (1.70)

15. Secondary Outcome: Visual Analog Scale - Language/Communication Score
Description: The Visual Analog Scale measures the severity of three specific behavioral symptoms as reported by the parent/caregiver: Language/Communication, Anxiety/Obsessive Compulsive Behaviors, and Aggression/Hyperactivity/Hyperarousal. Caregivers mark on a visual line measuring 10 cm with "worst behavior" at 0 cm and "best behavior" at 10 cm. For each behavior the caregiver is instructed to mark their impression of the behavior at baseline visit and again at the six-month visit. The calculated distance in cm between the marks drawn at the baseline and six-month visits thereby demonstrates whether each behavior improved, worsened, or stayed the same during the study, and by how much. Shown here is the mean distance in cm from the "worst behavior" side for the Language/Communication scale, at the six-month visit. The smaller the value, the worse the behavior. The range is minimum 0 cm to maximum 10 cm.
Time Frame: At six-month visit
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | Sertraline Liquid Placebo | Sertraline Active Medication
Number analyzed (Participants) | 21 | 25
centimeters | 5.53 (2.95) | 4.70 (2.73)

ADVERSE EVENTS:
Time Frame: From baseline to follow-up (6 months).
Arm/Group | Sertraline Liquid Placebo | Sertraline Active Medication
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/26 | 1/32
Other Adverse Events (participants affected / at risk) | 26/26 | 30/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sertraline Liquid Placebo (N=26) | Sertraline Active Medication (N=32)
Hospitalization for dehydration (Infections and infestations) | 0 (0) | 1 (1) — Hospitalization for dehydration secondary to viral infection.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sertraline Liquid Placebo (N=26) | Sertraline Active Medication (N=32)
Upper respiratory infection (Infections and infestations) | 19 (39) | 23 (48)
Diarrhea (Gastrointestinal disorders) | 15 (17) | 8 (11)
Hyperactivity (Psychiatric disorders) | 9 (13) | 12 (14)
Sleep disturbance (Psychiatric disorders) | 3 (3) | 10 (14)
Irritability/Aggression (Psychiatric disorders) | 10 (11) | 7 (9)
Fever (Infections and infestations) | 7 (8) | 6 (10)
Vomiting (Gastrointestinal disorders) | 3 (3) | 7 (9)
Gastroenteritis (Gastrointestinal disorders) | 5 (7) | 7 (7)
Otitis media (Infections and infestations) | 2 (2) | 5 (7) — Ear infection
Rash (Skin and subcutaneous tissue disorders) | 4 (6) | 1 (1)
Lethargy (Psychiatric disorders) | 4 (5) | 3 (3)
Tic (Nervous system disorders) | 0 (0) | 2 (4)
Constipation (Gastrointestinal disorders) | 3 (3) | 1 (2)
Seasonal allergies (Immune system disorders) | 2 (3) | 1 (1)
Decreased appetite (Gastrointestinal disorders) | 1 (1) | 3 (3)
Dilated pupils (Eye disorders) | 1 (2) | 0 (0)
Eye redness (Eye disorders) | 2 (2) | 0 (0)
Obsessive behaviors (Psychiatric disorders) | 2 (2) | 0 (0)
Self-injurious behavior (Psychiatric disorders) | 1 (2) | 1 (1)
Encopresis (Gastrointestinal disorders) | 0 (0) | 2 (2)
Increased stimming (Psychiatric disorders) | 1 (1) | 2 (2)
Mouthing/chewing objects (Psychiatric disorders) | 0 (0) | 2 (2)
Regression (Psychiatric disorders) | 0 (0) | 2 (2)
Teeth grinding (Psychiatric disorders) | 1 (1) | 2 (2)
Cut (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Enuresis (Renal and urinary disorders) | 1 (1) | 1 (1)
Excessive drooling (Nervous system disorders) | 1 (1) | 0 (0)
Hand Foot Mouth Disease (Infections and infestations) | 1 (1) | 0 (0)
Headaches (Nervous system disorders) | 1 (1) | 0 (0)
Increase in pica (Psychiatric disorders) | 1 (1) | 0 (0)
Itching (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Localized left leg swelling (Immune system disorders) | 1 (1) | 0 (0) — Localized left leg swelling following routine immunizations.
Gray matter heterotopia (Nervous system disorders) | 1 (1) | 0 (0) — Gray matter heterotopia near one of the ventricles noted on MRI during the course of the study.
PE tube surgery (Ear and labyrinth disorders) | 1 (1) | 0 (0) — Pressure equalizer tube surgery
Possible seizure/syncope (Nervous system disorders) | 1 (1) | 0 (0)
Separation anxiety (Psychiatric disorders) | 1 (1) | 1 (1)
Sprained ankle (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Staph infection (Infections and infestations) | 1 (1) | 0 (0)
Tuberous sclerosis (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) — Diagnosis was suspected prior to subject's enrollment in the trial but was confirmed during the course of trial participation.
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0)
Burned feet (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — Scalded skin on bottoms of both feet on hot water in bathtub, accidental burn.
Chicken pox (Infections and infestations) | 0 (0) | 1 (1)
Flu (Infections and infestations) | 0 (0) | 1 (1)
Gas (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hoarding (Psychiatric disorders) | 0 (0) | 1 (1)
Inappropriate laughing (Psychiatric disorders) | 0 (0) | 1 (1)
Inattention (Psychiatric disorders) | 0 (0) | 1 (1)
Increased frequency of bowel movements (Gastrointestinal disorders) | 0 (0) | 1 (1)
Tooth pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Not having minimum or maximum verbal or other developmental requirements to qualify for inclusion in this study. Sample size is small due to significant recruitment/retention challenges. Study power threshold was not met.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-06-15): https://cdn.clinicaltrials.gov/large-docs/99/NCT02385799/Prot_SAP_000.pdf